CLINICAL TRIAL: NCT00006903
Title: Phase II Study of Faslodex ? in Recurrent/Metastatic Endometrial Carcinoma
Brief Title: Fulvestrant in Treating Patients With Recurrent, Persistent, or Metastatic Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0188; NCI-2009-00581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068339; GOG-0188 (Other: NRG Oncology); GOG-0188 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Fulvestrant

ARMS (1):
- Treatment (fulvestrant) (Experimental): Patients receive fulvestrant intramuscularly on day 1. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Given intramuscularly
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238

SUMMARY:
This phase II trial is studying fulvestrant to see how well it works in treating patients with recurrent, persistent, or metastatic endometrial cancer. Estrogen can stimulate the growth of cancer cells. Hormone therapy using fulvestrant may fight cancer by blocking the uptake of estrogen by the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the probability of clinical response in estrogen receptor (ER)-positive vs ER-negative patients with recurrent, persistent, or metastatic endometrial cancer treated with fulvestrant.

II. Compare the relationship between response rate and intensity of receptor expression in patients treated with this drug.

III. Determine the frequency and intensity of toxicity of this drug in these patients.

OUTLINE:

Patients receive fulvestrant intramuscularly on day 1. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Criteria:

* Histologically confirmed recurrent, persistent, or metastatic endometrial cancer that is not curable with surgery or radiotherapy
* Estrogen receptor (ER) and progesterone receptor status known by immunohistochemistry

  * ER positive or negative allowed
* Measurable disease:

  * At least 1 target lesion not within a previously irradiated field OR irradiated target lesion with clear disease progression
  * At least 20 mm by conventional techniques, including palpation, x-ray, CT scan, MRI, OR at least 10 mm by spiral CT scan
* Performance status:

  * GOG 0-1
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm^3
  * Platelet count >= 100,000/mm^3
  * No prior bleeding diathesis (disseminated intravascular coagulation, clotting factor deficiency, or requirement for anticoagulants)
* Hepatic:

  * Bilirubin =< 1.5 times upper limit of normal (ULN)
  * SGOT =< 3 times ULN
  * Alkaline phosphatase =< 3 times ULN
* Renal:

  * Creatinine =< 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hypersensitivity to castor oil
* No other concurrent malignancy except nonmelanoma skin cancer
* No other prior malignancy within past 5 years
* No prior chemotherapy for persistent, recurrent, or metastatic endometrial cancer
* No more than 1 prior chemotherapy regimen for newly diagnosed endometrial cancer that has subsequently recurred
* At least 3 weeks since prior hormonal therapy and recovered
* At least 3 weeks since prior radiotherapy and recovered
* At least 3 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-08-30 (Actual); Primary Completion 2008-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan L Covens, Principal Investigator — NRG Oncology

RESULTS

PARTICIPANT FLOW:
Groups:
- Ineligible: Not eligible
- Estrogen Receptor Negative: Estrogen Receptor Negative, Faslodex® 250mg intramuscularly per month, minimum treatment period two cycles until disease progression or adverse effects prohibit further therapy
- Estrogen Receptor Positive: Estrogen Receptor Postive, Faslodex® 250mg intramuscularly per month, minimum treatment period two cycles until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Ineligible | Estrogen Receptor Negative | Estrogen Receptor Positive
Started | 10 | 24 | 33
Completed | 0 | 20 | 27
Not Completed | 10 | 4 | 6
Not completed — Still receiving treatment | 0 | 0 | 1
Not completed — Refused further treatment | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Patient never treated | 0 | 0 | 1
Not completed — Ineligible | 10 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Total number of eligible and treated participants by estrogen receptor status in metastatic tumor
Groups:
- Total: Total of all reporting groups
Arm/Group | Estrogen Receptor Negative | Estrogen Receptor Positive | Total
Number analyzed (Participants) | 23 | 30 | 53
Age, Customized [Mean (Standard Deviation); unit: years] | 62.9 (10.2) | 65.9 (10.4) | 64.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria Evaluated Every 8 Weeks
Description: Primary outcome measured according to RECIST v1.0 Best Response:
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart
  Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of nontarget lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required
  Stable Disease is any condition not meeting the above criteria.
  Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: Response was measured every other cycle (every 8 weeks) until disease progression is documented or adverse events preclude further treatment.
Population: Total number eligible and treated participants within groups defined by estrogen receptor status in metastatic tumor.
Measure: Number; unit: participants
Arm/Group | Estrogen Receptor Negative | Estrogen Receptor Positive
Number analyzed (Participants) | 23 | 30
participants
  Complete Response | 0 | 1
  Partial Response | 0 | 4
  Stable Disease | 4 | 9
  Disease Progression | 18 | 16
  Indeterminate | 1 | 0

2. Primary Outcome: Clinical Response by RECIST Criteria of Estrogen Receptor Expression
Description: Per response evaluation criteria in Solid Tumors Criteria (RECIST 1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >=30% decrease in the sum of the longest diameter of target lesions. Overall Response = CR+PR
Time Frame: Every other cycle (every 8 weeks) until disease progression is documented or adverse events preclude further treatment, assessed up to 100 months.
Population: Total number eligible and treated participants within groups defined by estrogen receptor status
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Receptor Negative | Estrogen Receptor Positive
Number analyzed (Participants) | 22 | 31
Participants
  Complete Response | 0 | 1
  Partial Response | 0 | 4
  Stable Disease | 4 | 9
  Increasing Disease | 17 | 17
  Not Evaluated | 1 | 0

3. Secondary Outcome: Number of Participants With Grade 3 or Greater Toxicity by Common Toxicity Criteria Version 3.0 That Were at Least Possibly Related to Study Drug.
Description: Adverse events at least possibly related to Fulvestrant using Common Terminology Criteria version 3.0 that were grade 3 or higher with the exception of the reported Grade 5. Grade 5 adverse events were reported regardless of attribution to study treatment.
Time Frame: During study treatment and up to 30 days after stopping study
Population: Eligible and evaluable patients.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5: Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Anemia | 1 | 1 | 0
  Fatigue | 1 | 0 | 0
  Gastrointestinal | 1 | 0 | 0
  Nausea | 3 | 0 | 0
  Vomiting | 1 | 0 | 0
  Diarrhea | 1 | 0 | 0
  Anorexia | 2 | 0 | 0
  Metabolic | 2 | 0 | 0
  Neurologic | 2 | 0 | 0
  Depression | 1 | 0 | 0
  Pain | 1 | 0 | 0
  Dyspnea | 1 | 0 | 0
  Thrombosis/embolism, regardless of attribution | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: Study treatment, and up to 30 days after stopping study treatment.
Description: The frequencies of maximum grade of serious adverse event or, for other adverse events, treatment-related adverse events by category or specific term occurring during treatment and up to 30 days after stopping the study treatment are reported.
  Other Adverse Events reported are Grade 2 or higher.
Groups:
- Faslodex: Faslodex® 250mg intramuscularly per month, minimum treatment period two cycles until disease progression or adverse effects prohibit further therapy.
  Includes both Estrogen Receptor Positive and Estrogen Receptor Negative participants.
Arm/Group | Faslodex
Serious Adverse Events (participants affected / at risk) | 11/53
Other Adverse Events (participants affected / at risk) | 28/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faslodex (N=53)
Death no ctcae term - disease progression (General disorders) | 1
Death no ctcae term - death nos (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Obstruction, gi - small bowel nos (Gastrointestinal disorders) | 1
Hemorrhage, gi - stomach (Vascular disorders) | 1
Hemorrhage/pulmonary - respiratory tract (Vascular disorders) | 1
Infection - other (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pain: abdominal pain nos (General disorders) | 1
Pain: pelvis (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faslodex (N=53)
Anemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 1
Auditory (Ear and labyrinth disorders) | 1
Constitutional (General disorders) | 3
Fatigue (General disorders) | 13
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1
Hot Flashes/Flushes (Endocrine disorders) | 6
Gastrointestinal (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 8
Infection/Fever (Infections and infestations) | 1
Metabolic (Metabolism and nutrition disorders) | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1
Neurologic (Nervous system disorders) | 3
Depression (Nervous system disorders) | 6
Ocular/Visual (Eye disorders) | 1
Pain (General disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Thrombosis/embolism (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
Accrual was discontinued after completion of the first stage of accrual due to lack of study drug activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No